CLINICAL TRIAL: NCT00001121
Title: Evaluation of Virologic, Immunologic, and Clinical Parameters of Participants in HIVNET 014 Who Become Infected With HIV-1
Brief Title: A Study to Monitor the Health of Participants in HIVNET 014 Who Become Infected With HIV-1
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: HIVNET 014A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections
Keywords: Placebos; AIDS Vaccines; Follow-Up Studies; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to evaluate the long-term consequences of HIV-1 infections that occurred in association with known, but discouraged, high-risk behaviors in persons who have received HIV candidate vaccines or placebo in HIVNET 014. Doctors need to look at how these patients respond to HIV infection in order to develop new HIV vaccines and other treatments for HIV and AIDS.

Patients who receive HIV vaccines are sometimes protected from HIV infection. More often, these patients become HIV-positive but experience a boost in their immune system that helps their bodies fight HIV. Doctors need to look at how these patients respond to HIV infection in order to develop new HIV vaccines and other treatments for HIV and AIDS.

DETAILED DESCRIPTION:
There are many possible outcomes of HIV-1 infection among persons who receive experimental HIV-1 vaccines. In the best-case scenario, these vaccines may prevent infection (sterilizing immunity). However, current viral vaccines are thought to limit, but not prevent, virus replication after infection. In the latter case, it is important to document the effect of the immune response on the disease course as reflected by viral load, the evolution of the viral quasi species, and clinical symptoms over time. Understanding the evolution of the immune response in vaccinees after subsequent exposure and HIV infection will potentially result in valuable information for the subsequent design of preventive and therapeutic vaccines. This will be studied here using HIVNET 014 participants at higher risk for HIV-1 infection.

Participants discontinue HIVNET 014 vaccinations upon confirmation of HIV-1 infection and are enrolled in this study. Participants undergo clinical and laboratory examinations every 3 months for the first year of follow-up and every 6 months for at least 4 years thereafter. Additionally, HIV-infected partners of HIVNET 014A participants undergo clinical and laboratory examination at enrollment, and may be asked to donate additional specimens at a later time. Study endpoints include various virologic, immunologic, and clinical parameters, such as viral load, cellular immune response, and virus phenotype and genotype.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Become infected with HIV while participating in HIVNET 014, or if they are an HIV-positive partner (sexual or needle-sharing) of a HIVNET 014A participant.
* Are able and willing to provide written informed consent.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a serious psychiatric or psychological disorder that would prevent them from completing the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, Study Chair; Susan Buchbinder, Study Chair; Haynes Sheppard, Study Chair
Locations (11):
- United States (11):
  - San Francisco Dept of Hlth / AIDS Office, San Francisco, California
  - Denver Dept of Public Health / HIVNET, Denver, Colorado
  - Univ of Illinois Chicago / Howard Brown Hlth Ctr, Chicago, Illinois
  - Howard Brown Health Ctr / HIVNET, Chicago, Illinois
  - Fenway Community Health Ctr / HIVNET, Boston, Massachusetts
  - New York Univ Med Ctr, New York, New York
  - New York Blood Ctr, The Bronx, New York
  - Univ of Pennsylvania / HIVNET, Philadelphia, Pennsylvania
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Miriam Hosp, Providence, Rhode Island
  - Univ of Washington, Seattle, Washington